## **Cover Page**

The Official Title: Effects of Preoperative Rehabilitation on Tendon

Healing, Bone Mineral Density, and Cartilage After ACLR and

**Patellar Dislocation** 

**NCT Number: 05924178** 

Date of the Document: 06/10/2025

## **Statistical Analysis Plan**

SPSS 21.0 statistical software was utilized for statistical analysis. When the test index was normal distribution, it was expressed as x±sd. If the detection indexes did not follow a normal distribution, they were described by the median (P25, P75). For normally distributed data, repeated measures analysis of variance was employed to assess changes across baseline, pre-ACLR, 3 months post-ACLR, 6 months post-ACLR, and 12 months post-ACLR, while the non-parametric Friedman test was used for non-normally distributed data. P<0.05 was considered statistically significant.